CLINICAL TRIAL: NCT01763034
Title: Limb Ischemic Preconditioning for Prevention of Contrast Media Induced Nephropathy in Diabetic Kidney Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Sirapat Poonvutikul, Cardiology unit, Ramathibodi Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: RAMA-CIN01
Record Dates: First submitted 2012-12-23; First posted 2013-01-08 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Serum Cystatin C Before and After Coronary Angiogram; Serum Creatinine Before and After Coronary Angiogram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- limb ischemia (Sham Comparator)
  Interventions: Procedure: limb ischemic preconditioning

INTERVENTIONS:
Procedure: limb ischemic preconditioning — use a simple blood pressure cuff inflate for 5 minutes and deflate for 5 minutes alternately in each arms total = 3 cycle in each arm

SUMMARY:
Contrast media induced nephropathy (CIN) is considered to be a serious complication in patient who underwent coronary angiogram (CAG). The pathogenesis of CIN does not well understood. The probable one is the contrast media makes the afferent vessel in glomeruli constrict and results in renal shut down. Limb ischemic preconditioning, a procedure that makes muscles become ischemic and adapt themselves to produce some cytokines for signaling the vessel more dilated. After the reperfusion, these cytokines are getting back to systemic circulation and effect the afferent vessel in glomeruli to become more dilated and prevent CIN.

ELIGIBILITY:
Inclusion Criteria:

* Documented diabetic kidney disease
* Elective coronary angiogram
* Glomerular filtration rate < 60 ml/min by Cockroft-Gault or Modification of Diet in Renal Disease or CKD-EPI

Exclusion Criteria:

* Refuse or reject to inform consented
* Hemodynamic compromise (Heart failure, need for intraaortic balloon pump)
* Expose to drug or chemical substances potentially to be a nephrotoxic agent with in 1 mo (Not include preexisting Angiotensin converting enzyme inhibitor or Angiotensin receptor blocker with stable serum creatinine)
* Documented or suspected of peripheral arterial disease, upper or lower limb
* Bleeding diathesis
* Contraindicated for coronary angiogram
* currently on renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
kidney injury before and after coronary angiogram. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Bangkok, Thailand